CLINICAL TRIAL: NCT00267163
Title: Brain Imaging and Mental Disorders of Aging Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IA0090; 9R01AG018487-06 (NIH)
Record Dates: First submitted 2005-12-16; First posted 2005-12-20 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-08

CONDITIONS: Cognition Disorders
Keywords: Alzheimer's disease; Mild Cognitive Impairment
MeSH Terms: conditions — Cognition Disorders; Alzheimer Disease; Cognitive Dysfunction | interventions — Donepezil

ARMS (2):
- 1. (Experimental)
  Interventions: Drug: donepezil
- 2. (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: donepezil
  Arms: 1.
Drug: Placebo
  Arms: 2.

SUMMARY:
The goal of this project is to determine if a cholinesterase inhibitor is more effective than placebo in delaying cognitive and brain functional decline in people at risk for Alzheimer's disease.

DETAILED DESCRIPTION:
Studies to date show that pictures of the brain using PET (positron emission tomography) scan measures predict memory decline in people with genetic risks for developing AD. They have also been shown to predict memory decline in people with mild memory complaints. These findings are consistent with other evidence that the changes of Alzheimer's Disease (AD) begin years before the doctor can confirm a diagnosis.

In this study, PET and genetic risk studies will be performed in people with mild memory complaints. A total of 138 participants (age 40 to 90 years) who are at risk for further memory decline will be enrolled. They will be randomized (like the flip of a coin) to one of two treatment groups, donepezil (a medication to treat mild AD) or placebo, and followed 18 months for evidence of future decline. Participants will receive magnetic resonance imaging (MRI) scans, PET scans, genetic risk assessment for Alzheimer's Disease, and neuropsychological assessments. Repeat brain imaging studies will be performed at the end of the 18-month treatment trial.

These procedures will allow researchers to explore how baseline brain function and genetic risk for AD onset influences brain metabolic rate and memory decline, and treatment outcome. Participants receiving donepezil are expected to show less evidence of decline than those receiving placebo. This project will expand a growing research program in early detection and prevention of AD, designed (1) to identify persons without memory complaints who are most likely to benefit from early intervention and (2) to provide an objective way to monitor the activity in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate in a 18 month clinical trial
* NIMH diagnostic criteria for age-associated memory impairment (AAMI)
* Age 40 to 90 years
* MMSE score between 24 and 30 (unless < 8 years of educational achievement)
* No significant cerebrovascular disease - modified Ischemic Score of < 4
* The following medications are allowed if stable for > 1 month: antidepressants (without anticholinergic effects) if not currently depressed and no history of major depression for 2 years; estrogen replacement therapy; thyroid replacement therapy as long as patient is euthyroid
* On entering the study, there must be a family member or potential caregiver available in case the patient develops cognitive impairment that interferes with independent study participation.
* Memory and verbal fluency cut-off scores increasing the probability of incipient dementia (Buschke-Fuld - 34; verbal fluency - 46 for letters, 7 for categories; Benton Visual Retention - 5)
* Adequate visual and auditory acuity to allow neuropsychological testing
* Screening laboratory tests and ECG without significant abnormalities that might interfere with the study

Exclusion Criteria:

* Diagnosis of possible or probable AD or any other dementia (e.g., vascular, Lewy body, frontotemporal)
* Evidence of neurologic or other physical illness that could produce cognitive deterioration, including Parkinson's disease; volunteers with a history of TIAs, carotid bruits, or lacunes on MRI scan will be excluded
* History of myocardial infarction within the previous year or unstable cardiac disease
* Uncontrolled hypertension, history of significant liver disease, clinically significant pulmonary disease, diabetes, or cancer
* Such current major psychiatric disorders as mania, according to DSMIV criteria, within the previous two years
* Current diagnosis or history of alcoholism or drug dependence
* Evidence of untreated depression
* Use of any of the following drugs: centrally active beta-blockers, narcotics, clonidine, anti-Parkinsonian medications, antipsychotics, benzodiazepines, systemic corticosteroids, medications with significant cholinergic or anticholinergic effects, anti-convulsants, or warfarin; vitamins other than the standard multivitamin supplement, ginkgo biloba, and any nutraceuticals will not be allowed; once enrolled in the study, occasional chloral hydrate use will be allowed, but discouraged, for insomnia
* Use of any investigational drugs within the previous month or longer, depending on drug half-life
* Contraindication for MRI scan (e.g., metal in body, claustrophobia)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2000-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Changes in cognition and brain metabolism measured by PET and MRI scans, and neuropsychological testing | at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary W. Small, MD, Principal Investigator — University of California, Los Angeles, Neuropsychiatric Institute
Locations (1):
- UCLA, The Semel Institute for Neuroscience and Human Behavior, Los Angeles, California, United States

REFERENCES:
- [Background] Small SA, Stern Y, Tang M, Mayeux R. Selective decline in memory function among healthy elderly. Neurology. 1999 Apr 22;52(7):1392-6. doi: 10.1212/wnl.52.7.1392. PMID 10227623
- [Background] Small GW, Chen ST, Komo S, Ercoli L, Bookheimer S, Miller K, Lavretsky H, Saxena S, Kaplan A, Dorsey D, Scott WK, Saunders AM, Haines JL, Roses AD, Pericak-Vance MA. Memory self-appraisal in middle-aged and older adults with the apolipoprotein E-4 allele. Am J Psychiatry. 1999 Jul;156(7):1035-8. doi: 10.1176/ajp.156.7.1035. PMID 10401448
- [Background] Ercoli LM, Siddarth P, Dunkin JJ, Bramen J, Small GW. MMSE items predict cognitive decline in persons with genetic risk for Alzheimer's disease. J Geriatr Psychiatry Neurol. 2003 Jun;16(2):67-73. doi: 10.1177/0891988703016002001. PMID 12801154
- [Background] Silverman DH, Small GW, Chang CY, Lu CS, Kung De Aburto MA, Chen W, Czernin J, Rapoport SI, Pietrini P, Alexander GE, Schapiro MB, Jagust WJ, Hoffman JM, Welsh-Bohmer KA, Alavi A, Clark CM, Salmon E, de Leon MJ, Mielke R, Cummings JL, Kowell AP, Gambhir SS, Hoh CK, Phelps ME. Positron emission tomography in evaluation of dementia: Regional brain metabolism and long-term outcome. JAMA. 2001 Nov 7;286(17):2120-7. doi: 10.1001/jama.286.17.2120. PMID 11694153
- [Background] Small GW, Ercoli LM, Silverman DH, Huang SC, Komo S, Bookheimer SY, Lavretsky H, Miller K, Siddarth P, Rasgon NL, Mazziotta JC, Saxena S, Wu HM, Mega MS, Cummings JL, Saunders AM, Pericak-Vance MA, Roses AD, Barrio JR, Phelps ME. Cerebral metabolic and cognitive decline in persons at genetic risk for Alzheimer's disease. Proc Natl Acad Sci U S A. 2000 May 23;97(11):6037-42. doi: 10.1073/pnas.090106797. PMID 10811879